CLINICAL TRIAL: NCT02874690
Title: Title: Eye Tracking as a Predictor of Methylphenidate Response in Autism With Co-morbid Attention Deficit Hyperactivity Disorder
Brief Title: Eye Tracking as a Predictor of Methylphenidate Response in Autism With ADHD
Acronym: SAT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015-4401
Record Dates: First submitted 2016-03-04; First posted 2016-08-22 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo pill received
  Interventions: Drug: Placebo
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — single dose methylphenidate; 0.3mg/kg, up to 20mg, rounded to the nearest 2.5mg
  Arms: Methylphenidate
Drug: Placebo — Placebo pill identical in appearance to methylphenidate
  Arms: Placebo

SUMMARY:
The overall goal of this research is to use neurophysiological measures to profile strengths and deficits for Attention Deficit Hyperactivity Disorder co-morbidity in Autism Spectrum Disorder to clarify diagnosis and to predict treatment response.

DETAILED DESCRIPTION:
The project "Eye Tracking as a Predictor of Methylphenidate (MPH) Response in Low Functioning Autism Spectrum Disorders (ASD) with comorbid ADHD" will investigate the role of a non-invasive neurophysiological biomarker in an underserved population to clarify diagnosis and guide treatment decisions. Specifically, we will modify an existing eye tracking paradigm that discriminates between ADHD and typical youth, for use in an ASD cohort with (ASD+) and without an ADHD comorbidity. A case-control design (Aim 1) will lead into a randomized placebo controlled trial of MPH in children with ASD with comorbid ADHD (Aim 2). We hypothesize that children with ASD+ will demonstrate specific abnormalities in microsaccades, eye blink frequency, and pupil dilatation on continuous performance testing that will predict MPH treatment response on standardized clinical outcomes for ADHD. As a secondary measure, we will also perform a brief electrophysiological measure, short interval cortical inhibition (SICI), as measured by paired pulse transcranial magnetic stimulation (TMS). We have extensively investigated this measure as a robust predictor of ADHD diagnosis and symptom severity in ADHD and typical youth. We anticipate this personalized medicine-based approach to clarify ADHD co-occurrence in ASD will result in a novel neurophysiological biomarker will enhance diagnostic reliability and better match appropriate pharmacotherapy in a highly complex neurodevelopmental disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual 5 (DSM-V) diagnosis of Autism Spectrum Disorder (ASD) not otherwise specified (NOS) based on a semi-structured review of Diagnostic and Statistical Manual 5 (DSM-V) criteria and mental status examination as well as a a complete systematic patient interview utilizing the Autism Diagnostic Observation Schedule (ADOS)
* Males and females ages 8-21 years.
* Subjects must not be taking any psychotropic drugs affecting glutamate neurotransmission (riluzole, memantine, acamprosate, topiramate, amantadine, among others) which may interfere with TMS recording. If patient is on a home psychostimulants medication this will be held on the day of testing. Subjects may not be taking more than two psychotropic drugs. Dosing of all concomitant psychotropic drugs targeting core social and/or communication impairment must be stable for four weeks prior to randomization. Dosing of all concomitant psychotropic drugs targeting other features associated with ASD (insomnia, inattention, hyperactivity, anxiety, irritability among others) must be stable for two weeks (with the exception of four weeks for fluoxetine) prior to randomization.
* Stable seizure disorder (no seizures in 6 months prior to enrollment; on same anticonvulsant dose > 60 days or )
* Able to participate in neurophysiological testing including Electroencephalogram (EEG) and Transcranial Magnetic Stimulation (TMS) portions of the experiment based on patient comfort and examiner judgement
* Legal guardian has provided written informed consent and the subject has provided written informed assent. Expectation that a majority of subjects will be able to assent but the potential for the younger children and/or those that are cognitively impaired will not be able to assent.

Exclusion Criteria:

* Subjects exhibiting significant disruptive, aggressive, self-injurious, or sexually inappropriate behavior will not be eligible for enrollment
* Presence of current Diagnostic and Statistical Manual 5 (DSM-V) psychiatric disorders that may require alternative pharmacotherapy or different treatment including psychotic disorders, major affective disorders, obsessive-compulsive disorder, panic disorder, or substance related disorders.
* Presence of any medical condition that would make treatment with methylphenidate (MPH) less safe. Subjects with significant cardiac, hepatic, or renal disease will be excluded due to concerns about pharmacokinetic alterations or adverse effects. Because of the unknown effects of methylphenidate (MPH) on the developing human fetus, females of childbearing potential will be given a urine pregnancy test and required to use a suitable form of birth control during the study. A positive pregnancy test result excludes the subject.
* Presence of any other condition that would make the participants unable to comply with the requirements of the study for any reason.
* Prohibited Concomitant Medications: Methylphenidate is primarily excreted by the kidneys and has few known pharmacokinetic drug interactions. The following medications are not allowed due to the potential for a pharmacodynamic interaction: monoamine oxidase inhibitors or atomoxetine.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Change in Eye-Tracking: Microsaccades and pupil size using Tobii eye tracker | Pre-dose; Approximately 90 minutes post-dose of methylphenidate
  Eye tracking offers a window into a "hardwired" circuit into the brain in a patient population that may not easily tolerate more invasive diagnostic procedures.

SECONDARY OUTCOMES:
Change in Short Interval IntraCortical Inhibition (SICI) using Transcranial Magnetic Stimulation (TMS) | Pre-dose; Approximately 90 minutes post-dose of methylphenidate
  SICI is a TMS measure of the efficiency of inhibitory interneurons in the primary motor cortex.
Change in Resting State Electroencephalogram (EEG) | Pre-dose; Approximately 90 minutes post-dose of methylphenidate
  EEG will be used to assess the electrophysiologic aspects of behavioral computerized testing, behavior, or motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Pedapati, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT02874690/Prot_SAP_000.pdf